CLINICAL TRIAL: NCT06789484
Title: Recovery of a Probiotic in Term Newborns - a Randomized, Double-blinded, Placebo-controlled Proof-of-concept Study
Brief Title: Characterization of the Gastrointestinal Microbiota in Newborn Infants
Acronym: BABIES I
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Chr Hansen (Industry)
Responsible Party: Principal Investigator, Andreas Munk Petersen, Professor Andreas Munk Petersen, MD, PhD, DMSc, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HND-IN-056; H-24073138 (Other: Ethics Committee Case number)
Record Dates: First submitted 2025-01-06; First posted 2025-01-23 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Healthy Infants
Keywords: Infant; Gastrointestinal Microbiome; Diet, Food, and Nutrition
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A randomized, controlled trial of healthy term in newborns with a 4-week intervention period from birth to 28 days of life followed by a 2-week follow-up period
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): Probiotic Dietary supplement
  Interventions: Other: Probiotic
- Placebo (Placebo Comparator): Identical looking placebo consisting of maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Other: Probiotic — Given daily from enrollement to 28 days of life
  Arms: Probiotic
Dietary Supplement: Placebo — Given daily from enrollement to 28 days of life
  Arms: Placebo

SUMMARY:
The BABIES study is a single-center, randomized, double-blinded, placebo-controlled study in newborns with a 4-week intervention period from birth to 28 days of life followed by a 2-week follow-up period (Figure 1). The study will evaluate the seeding ability of supplementation with a probiotic strain.

The aim is to investigate the recovery and engraftment of the probiotic strain in infant fecal samples after 4 weeks supplementation using a strain specific quantitative Polymerase Chain Reaction (qPCR).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria for the pregnant person:

  1. Healthy pregnant person in gestational week 36+0-38+0
  2. Age ≥ 18 years
  3. Normal singleton pregnancy
  4. Ability to read and speak Danish
  5. Normal ultrasound scan of the fetus at gestational age 19-20 weeks
  6. Plan to exclusively breastfeed
  7. Provided voluntary written informed consent.
* Inclusions Criteria for the newborn:

  1. Born at full-term ≥37+0
  2. Birth weight above 2500 g
  3. APGAR score of at least 7 within the first 5 min of life.

     Exclusion Criteria:
* Exclusion Criteria for the pregnant person:

  1. Pregnancy at over 38+0 weeks' gestation at recruitment
  2. Multiple pregnancy
  3. Pregnancy with any fetal abnormality
  4. Alcohol or drug abuse
  5. Plan to give birth at other hospitals than Copenhagen University Hospital Hvidovre
  6. Any contraindications for breastfeeding.

Exclusion Criteria for the newborn :

1. Congenital disorders that could affect their safety or the study outcome
2. Admission to Neonatal Intensive Care Unit for more than 24 hours
3. Participation in another clinical intervention study which can interfere with this probiotic intervention
4. No other probiotics than the study product.

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovery of the probiotic strain in newborn/infant fecal samples | Birth (first stool after meconium), 2 weeks, 4 weeks, and 6 weeks
  Abundance of the probiotic strain in newborn/infant fecal samples measured by quantitative PCR.

SECONDARY OUTCOMES:
Infant fecal pH | Birth (first stool after meconium), 2 weeks, 4 weeks, and 6 weeks
  Changes in Fecal pH measured in fecal water from fecal samples.
Total abundance of bifidobacteria | Birth (first stool after meconium), 2 weeks, 4 weeks, and 6 weeks
  Abundance of fecal bifidobacteria measured by quantitative PCR
Infant fecal short chain fatty acids (SCFA) | Birth (first stool after meconium), 2 weeks, 4 weeks, and 6 weeks
  Changes in SCFA production as measured by targeted metabolomics

OTHER OUTCOMES:
Infant gut metabolome | Birth (first stool after meconium), 2 weeks, 4 weeks, and 6 weeks
  Characterization and changes in the Infant fecal metabolome as assessed by targeted and untargeted metabolomics in infant fecal samples
Infant gut microbiome composition | Birth (first stool after meconium), 2 weeks, 4 weeks, and 6 weeks
  Changes in gut microbiome composition analyzed by DNA/RNA sequencing of fecal samples
Infant blood metabolome | 4 weeks
  Newborn blood metabolome as assessed by targeted and untargeted metabolomics from dried blood spots
Infant bowel habits frequency | Daily (0-6 weeks of age)
  Changes in bowel habits as measured by daily stool frequency.
Infant bowel habits stool consistency | Daily from 0-6 weeks of age
  Changes in bowel habits as measured by stool consistency. The consistency will be assessed by a modified diapered infant stool scale.
Infant growth, weight | Birth, 4 weeks, 6 weeks of age.
  Infant weight in kilograms will be aggregated to determine infant growth status.
Infant crying and fussing | Daily (0-6 weeks of age)
  Measured as frequency and duration (hours/minutes per day) of crying and fussing
Pregnant person fecal microbiota composition | 36+0-38+0 GA weeks
  Gut microbiome composition analyzed by DNA/RNA sequencing of fecal samples
Pregnant person blood metabolome | 36+0-38+0 GA weeks
  Characterization of the pregnant person blood metabolome as assessed by targeted and untargeted metabolomics from dried blood spots
Infant growth, length | Birth, 4 weeks, 6 weeks of age.
  Infant length in centimeters will be aggregated to determine infant growth status.
Infant growth, head circumference | Birth, 4 weeks, 6 weeks of age.
  Infant head circumference in centimeters will be aggregated to determine infant growth status.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Munk Petersen, MD, PhD, DMSc, Principal Investigator — Center for Klinisk Mikrobiom Forskning, Gastroenheden og Klinisk Mikrobiologisk Afdeling, Hvidovre Hospital
Locations (1):
- Center for Klinisk Mikrobiom Forskning, Gastroenheden og Klinisk Mikrobiologisk Afdeling, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No